CLINICAL TRIAL: NCT04097236
Title: Diagnostic Performance of the Ultrasound Examination of the Antrum to Detect a Full Stomach According to the Position of the Patient
Brief Title: Body Position and Ultrasound Examination of the Gastric Antrum
Acronym: POSIGAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL19_0244; 2019-A01333-54 (Other: ID-RCB)
Record Dates: First submitted 2019-05-15; First posted 2019-09-20 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Aspiration of Gastric Contents
MeSH Terms: conditions — Respiratory Aspiration of Gastric Contents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 45° semirecumbent position (Active Comparator)
  Interventions: Other: Qualitative and quantitative assessment of gastric content volume with bed elevation
- No elevation of the upper section of the bed (Active Comparator)
  Interventions: Other: Qualitative and quantitative assessment of gastric content volume without bed elevation

INTERVENTIONS:
Other: Qualitative and quantitative assessment of gastric content volume with bed elevation — Ultrasound examination of the gastric antrum are performed 3 minutes after the ingestion of a volume of water (either 0, 50, 100, 150, or 200 milliliters (ml), determined by randomization). The procedure is repeated three times (three different volumes, the same volumes for each session with randomized order for each session).
  Arms: 45° semirecumbent position
Other: Qualitative and quantitative assessment of gastric content volume without bed elevation — Ultrasound examination of the gastric antrum are performed 3 minutes after the ingestion of a volume of water (either 0, 50, 100, 150, or 200 milliliters (ml), determined by randomization). The procedure is repeated three times (three different volumes, the same volumes for each session with randomized order for each session).
  Arms: No elevation of the upper section of the bed

SUMMARY:
Pulmonary aspiration of gastric contents is a complication causing significant morbidity and mortality related to anesthesia. Ultrasound examination of the gastric antrum allows the detection of preoperative gastric contents contributing to the preoperative assessment of pulmonary aspiration risk. In particular, this examination is based on the qualitative analysis of gastric contents performed in the supine and in the right lateral decubitus, using a qualitative score which makes it possible to discriminate a low liquid content of a large liquid volume. This score has been described in patients and volunteers installed on a bed without elevation of the upper section of the bed. However, in several studies, this qualitative score has been achieved in the 45° semirecumbent position, which may have affected the diagnostic performance of the examination thus performed, as suggested by the results of a study recently conducted by the investigating team. This study therefore aims to compare the diagnostic performance of the qualitative analysis of the gastric antrum performed in the supine and the right lateral decubitus for the diagnosis of gastric volumes higher than 50 ml and 100 ml, according to the bed angle: 45 ° elevation or no elevation of the upper section of the bed.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years old or older
* Last consumption of solids at least 6 hours before the start of the study, last consumption of clear fluids at least 2 hours before the start of the study
* Informed consent must have been signed.
* No significant medical history (American Society of Anesthesiologists (ASA) class 1)

Exclusion Criteria:

* Adult unable to give informed consent
* Previous gastrointestinal surgery
* Medication affecting gastric motility
* Digestive diseases, gastroparesis, diabetes mellitus with insulin
* Pregnancy or breastfeeding
* Obesity (Body Mass Index (BMI) ≥ 30 kilograms/meter² (kg/m²))

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2021-09-06 (Actual); Study Completion 2021-09-06 (Actual)

PRIMARY OUTCOMES:
Calculation of the sensitivity | 3 minutes
  Diagnostic performance of the qualitative examination of the gastric antrum in the 45° semirecumbent position.

SECONDARY OUTCOMES:
Calculation of the specificity | 3 minutes
  Diagnostic performance of the qualitative examination of the gastric antrum in full supine/right lateral decubitus position.
  The diagnostic performance will be calculated according to the results of the qualitative assessments performed 3 minutes after the ingestion of water (either 0, 50, 100, 150 or 200 milliliters (ml)) by the volunteers.
Calculation of the positive predictive value, | 3 minutes
  Diagnostic performance of the qualitative examination of the gastric antrum in full supine/right lateral decubitus position. The diagnostic performance will be calculated according to the results of the qualitative assessments performed 3 minutes after the ingestion of water (either 0, 50, 100, 150 or 200 milliliters (ml)) by the volunteers.
Calculation of the negative predictive value | 3 minutes
  Diagnostic performance of the qualitative examination of the gastric antrum in full supine/right lateral decubitus position. The diagnostic performance will be calculated according to the results of the qualitative assessments performed 3 minutes after the ingestion of water (either 0, 50, 100, 150 or 200 milliliters (ml)) by the volunteers.
Calculation of the positive and negative likelihood ratio. | 3 minutes
  Diagnostic performance of the qualitative examination of the gastric antrum in full supine/right lateral decubitus position. The diagnostic performance will be calculated according to the results of the qualitative assessments performed 3 minutes after the ingestion of water (either 0, 50, 100, 150 or 200 milliliters (ml)) by the volunteers.
Diagnostic performance of the qualitative examination of the gastric antrum for the detection of gastric fluid volume ≥ 0.8 milliliters/kilogram (ml/kg) in the full supine and right lateral decubitus position and in the 45° semirecumbent position | 3 minutes
  Calculation of the sensitivity. The diagnostic performance will be calculated according to the results of the qualitative assessments performed 3 minutes after the ingestion of water (either 0, 50, 100, 150 or 200 milliliters (ml)) by the volunteers
Diagnostic performance of the qualitative examination of the gastric antrum for the detection of gastric fluid volume ≥ 0.8 milliliters/kilogram (ml/kg) in the full supine and right lateral decubitus position and in the 45° semirecumbent position | 3 minutes
  Calculation of the specificity The diagnostic performance will be calculated according to the results of the qualitative assessments performed 3 minutes after the ingestion of water (either 0, 50, 100, 150 or 200 milliliters (ml)) by the volunteers
Diagnostic performance of the qualitative examination of the gastric antrum for the detection of gastric fluid volume ≥ 0.8 milliliters/kilogram (ml/kg) in the full supine and right lateral decubitus position and in the 45° semirecumbent position | 3 minutes
  Calculation of the positive predictive value negative The diagnostic performance will be calculated according to the results of the qualitative assessments performed 3 minutes after the ingestion of water (either 0, 50, 100, 150 or 200 milliliters (ml)) by the volunteers
Diagnostic performance of the qualitative examination of the gastric antrum for the detection of gastric fluid volume ≥ 0.8 milliliters/kilogram (ml/kg) in the full supine and right lateral decubitus position and in the 45° semirecumbent position | 3 minutes
  Calculation of the negative predictive value. The diagnostic performance will be calculated according to the results of the qualitative assessments performed 3 minutes after the ingestion of water (either 0, 50, 100, 150 or 200 milliliters (ml)) by the volunteers
Diagnostic performance of the qualitative examination of the gastric antrum for the detection of gastric fluid volume ≥ 0.8 milliliters/kilogram (ml/kg) in the full supine and right lateral decubitus position and in the 45° semirecumbent position | 3 minutes
  Calculation of the positive and negative likelihood ratio. The diagnostic performance will be calculated according to the results of the qualitative assessments performed 3 minutes after the ingestion of water (either 0, 50, 100, 150 or 200 milliliters (ml)) by the volunteers
Cut-off value for antral area measured in the supine position (semirecumbent or full supine position) associated with the best diagnostic performance for the detection of a gastric volume ≥1.5 milliliters/kilogram (ml/kg). | 3 minutes
  The cut-off value will be calculated according to the results of the measurements performed 3 minutes after the ingestion of water (either 0, 50, 100, 150 or 200 milliliters (ml)) by the volunteers
Diagnostic performance of the qualitative examination of the gastric antrum in the semirecumbent position without bed elevation | 3 minutes
  Calculation of the sensitivity. The diagnostic performance will be calculated according to the results of the qualitative and quantitative assessments performed 3 minutes after the ingestion of water (either 0, 50, 100, 150 or 200 milliliters (ml)) by the volunteers
Diagnostic performance of the qualitative examination of the gastric antrum in the semirecumbent position without bed elevation | 3 minutes
  Calculation of the specificity. The diagnostic performance will be calculated according to the results of the qualitative and quantitative assessments performed 3 minutes after the ingestion of water (either 0, 50, 100, 150 or 200 milliliters (ml)) by the volunteers
Diagnostic performance of the qualitative examination of the gastric antrum in the semirecumbent position without bed elevation | 3 minutes
  Calculation of the positive predictive value. The diagnostic performance will be calculated according to the results of the qualitative and quantitative assessments performed 3 minutes after the ingestion of water (either 0, 50, 100, 150 or 200 milliliters (ml)) by the volunteers
Diagnostic performance of the qualitative examination of the gastric antrum in the semirecumbent position without bed elevation | 3 minutes
  Calculation of the negative predictive value. The diagnostic performance will be calculated according to the results of the qualitative and quantitative assessments performed 3 minutes after the ingestion of water (either 0, 50, 100, 150 or 200 milliliters (ml)) by the volunteers
Diagnostic performance of the qualitative examination of the gastric antrum in the semirecumbent position without bed elevation | 3 minutes
  Calculation of the positive and negative likelihood ratio. The diagnostic performance will be calculated according to the results of the qualitative and quantitative assessments performed 3 minutes after the ingestion of water (either 0, 50, 100, 150 or 200 milliliters (ml)) by the volunteers
Mathematical model for the calculation of the gastric fluid volume | 3 minutes
  Multiple linear regression including the antral surface measured in right lateral decubitus and the age, height, weight of the volunteer. The mathematical model will be built according to the results of the measurements performed 3 minutes after the ingestion of water (either 0, 50, 100, 150 or 200 milliliters (ml)) by the volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Barnoud, Dr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Bron, France

REFERENCES:
- [Background] Bouvet L, Cordoval J, Barnoud S, Berlier J, Desgranges FP, Chassard D. Diagnostic performance of qualitative ultrasound assessment for the interpretation of point-of-care gastric ultrasound to detect high gastric fluid volume: A prospective randomized crossover study. J Clin Anesth. 2022 Oct;81:110919. doi: 10.1016/j.jclinane.2022.110919. Epub 2022 Jul 2. PMID 35792453